CLINICAL TRIAL: NCT03060616
Title: Validation of Hemorrhoidal Bleeding Score
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: SCORE_SG-hémorroide
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Hemorrhoid Bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The principal manifestation of hemorrhoidal disease is bleeding; however the severity evaluation is today based on prolapsus (Goligher classification) and bleeding factor is not included.

Even if there was some rare score including bleeding in literature , none of them were validated.

The aim of the study is first validation of bleeding score .

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* consulting for hemorroidal bleeding
* accept to participate

Exclusion Criteria:

* paraplegic or hemiplegic patient
* Misunderstanding of the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: every patient consulting for hemorrhoidal bleeding
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
assessment of bleeding score | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Hélène BEAUSSIER, Pharm-D, Study Director — CRC
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No